CLINICAL TRIAL: NCT05224206
Title: Neural Mechanisms of Intermittent Theta Burst Stimulation in the Core Depression Network
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Royal Ottawa Mental Health Centre (Other)
Responsible Party: Principal Investigator, Sara Tremblay, Scientist, The Royal Ottawa Mental Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021013
Record Dates: First submitted 2021-10-13; First posted 2022-02-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Major Depressive Disorder
Keywords: iTBS; rTMS; positron emission tomography
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be divided in two main parts. In Part I, we will use a randomized cross-over double-blinded design. The order of the iTBS conditions (active vs. sham) will be counterbalanced across participants. In part II, participants will receive a 6-week daily iTBS open-label treatment. Participants and research team members performing iTBS and analyses will be blind to the stimulation condition for Part I of the study. The order of the conditions will be determined by a separate research team member that will not be performing iTBS or analyses. Participants will be told that there is a sham condition, for Part I of the trial. The master randomization list was created by a scientist of the research centre that is not involved in the research project.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham iTBS/Active iTBS (Sham Comparator): Intermittent Theta Burst Stimulation (iTBS) or realistic sham iTBS will be applied to the left DLPFC. Both sessions will be one week apart.
  Interventions: Device: Theta burst stimulation
- Active iTBS (Active Comparator): Intermittent Theta Burst Stimulation (iTBS) will be applied to the left DLPFC. Participants will receive daily sessions (on weekdays) for 6 weeks.
  Interventions: Device: Theta burst stimulation

INTERVENTIONS:
Device: Theta burst stimulation — Cool B65 active/placebo coil (left DLPFC) with X100 MagPro rTMS Device (Magventure A/S, Farum, Denmark)
  Arms: Sham iTBS/Active iTBS
Device: Theta burst stimulation — Cool B70 coil (left DLPFC), with X100 MagPro rTMS Device (Magventure A/S, Farum, Denmark)
  Arms: Active iTBS

SUMMARY:
Repetitive Transcranial magnetic stimulation (TMS) uses magnetic fields to modulate brain activity. A novel form of repetitive TMS (rTMS), intermittent theta burst stimulation (iTBS), has emerged as a promising new treatment for depression. This technique may be advantageous due to its very short duration and potentially stronger effect on brain activity in comparison with standard rTMS. However, the exact effect of iTBS on the activity of the brain in clinical populations remains poorly understood. This project aims to improve understanding of the mechanisms of action of iTBS by comparing its neuronal effect to sham treatment in 22 individuals with a diagnosis of major depressive episode, using positron emission tomography (PET) and magnetic resonance imaging (MRI) in a double-blind cross-over experiment, followed by a 6-week daily treatment course of iTBS.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a Health Canada approved treatment for major depression. Typical clinical rTMS treatment is delivered on the left dorsolateral prefrontal cortex (DLPFC) at a 10 Hz frequency for 30-45 minutes to increase cortical excitability which will outlast the duration of stimulation. The treatment involves daily sessions that are applied over a four to six-week period. Intermittent theta burst stimulation (iTBS) is a novel refinement of conventional rTMS. iTBS consists of bursts of 3 stimulations at 50 Hz at theta frequency (5 Hz). However, instead of 30-min treatment sessions, iTBS has comparable clinical efficacy with only 3 minutes treatment sessions. Because iTBS is a novel technique, much of its effects on the brain are currently unknown. However, since it is a modified rTMS protocol, it is assumed that its neuronal effects are comparable.

Therapeutic effects of rTMS are thought to be related to its effects on the subgenual anterior cingulate cortex (sgACC; Broadman area 25). In depression, metabolic activity of the sgACC is increased (measured as increase of 18F-labeled fluorodeoxyglucose ([18F]FDG) uptake with positron emission tomography (PET)). Importantly, the metabolic activity of the sgACC appears to be a general marker for treatment response, e.g. [18F]FDG uptake is decreased in response to antidepressant medications or deep brain stimulation. In addition to resting state functional MRI, diffusion weighted imaging has been used to study TMS targets, but this technique has never been used for testing targets for treating depression.

Currently, the system level mechanisms of action of iTBS in depression patients are completely unexplored. Based on prior research the investigators hypothesize that 1) a single session of iTBS will decrease [18F]FDG uptake in the sgACC and 2) the magnitude of decrease is related to the connectivity between the target site and the sgACC. This study will establish the system level mechanisms of action of iTBS, paving a way to improve clinical treatment. This study will also develop connectivity measures that can be used to improve iTBS targeting (i.e. choose iTBS target based on sgACC connectivity) and predict treatment response (i.e. predict iTBS treatment response in patients based on sgACC connectivity).

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 to 55 years of age
* Mini-International Neuropsychiatric Interview-confirmed diagnosis of MDD, as a single or recurring episode
* Symptoms of MDD have not improved after ≥ 1 but ≤ 7 adequate dose(s) of antidepressant trial(s) in the current depressive episode
* A baseline score of ≥ 15 on the 17-item Hamilton Rating Scale for Depression (HRSD-17)
* Have received a stable antidepressant regimen for at least four weeks prior to entering trial
* Are voluntary and competent to consent to study
* Can speak and read English

Exclusion Criteria:

* Current or past (< 3 months) substance (including nicotine) or alcohol abuse/dependence, as defined in DSM-5 criteria
* Positive urine test for illegal substances, cannabis, or cotinine
* Suicide attempt in the past three months and/or active suicidal intent
* Pregnancy (confirmed by urine test) and/or lactation
* Psychotic features in the current episode
* Any comorbid mental health disorders (including, but not limited to lifetime history of psychotic disorders, OCD, PTSD and/or bipolar I or II disorder) with the exception of anxiety/panic disorders and ADHD
* Significant unstable medical or neurologic illness confirmed by medical history and blood test at baseline (e.g. uncontrolled diabetes, or renal dysfunction)
* Organic cause to the depressive symptoms (e.g. thyroid dysfunctions), as ruled out by the referring physician
* Contraindication for TMS (e.g., personal history of epilepsy or convulsion, metallic head implant, pacemaker)
* Contraindication for MRI (e.g. metallic implant, claustrophobia)
* Have undergone a prior PET or SPECT research study
* ECT or rTMS treatment in the current depressive episode
* Benzodiazepine use
* Have a body mass index (BMI) higher then 35 or lower then 18
* Any other condition that, in the opinion of the investigators, would adversely affect the participant's ability to complete the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Neural mechanisms of iTBS measured by [18F]FDG uptake in the sgACC | 40 minutes after iTBS
  The primary outcome measure for Part I is the change in [18F]FDG uptake in the sgACC after iTBS.
Neuroimaging predictors of iTBS response to treatment - primary measures | 6 weeks
  The primary clinical outcome measures will be response to treatment and remission. Response to treatment will be defined as at least a 50% reduction in pre-treatment symptoms severity as measured by the mean HRSD-17 score at week 6. Remission will be defined as a HRSD-17 score lower or equal to 7 at week 6.

SECONDARY OUTCOMES:
Neuroimaging predictors of iTBS response to treatment - QIDS-SR16 | 6 weeks
  For secondary analyses, improvement in symptoms will be defined as the percentage of change of symptoms at week 6 in comparison with pre-treatment symptoms severity. Response to treatment will be defined as a 50% reduction in pre-treatment symptoms severity as measured by the mean of the Quick Inventory of Depressive Symptomatology (16-item) (Self-Report) (QIDS-SR16). Remission will be defined as a QIDS-SR score ≤ 6.
Neuroimaging predictors of iTBS response to treatment - Beck Anxiety Inventory (BAI) | 6 week
  For secondary analyses, improvement in symptoms will be defined as the percentage of change of symptoms at week 6 in comparison with pre-treatment symptoms severity. Response to treatment will be defined as a 50% reduction in pre-treatment symptoms severity. The Beck Anxiety Inventory (BAI) will be used to assess severity of patient anxiety. It is a structured 21-item self-report measure using a likert scale of 0-3. A total score of 0 - 7 is interpreted as a "Minimal" level of anxiety; 8 - 15 as "Mild"; 16 - 25 as "Moderate", and; 26 - 63 as "Severe".
Neuroimaging predictors of iTBS response to treatment - Quality of life (Q-LES-Q-SF) | 6 week
  For secondary analyses, improvement in symptoms will be defined as the percentage of change of symptoms at week 6 in comparison with pre-treatment symptoms severity. Response to treatment will be defined as a 50% reduction in pre-treatment symptoms severity. The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) will be used to assess response to iTBS treatment. The Q-LES-Q-SF is used to obtain sensitive measures of the degree of enjoyment and satisfaction experienced by subjects in various areas of daily functioning. It's a structured 16-item self-report measure where items are scored on a 5-point Likert scale, from Very Poor to Very Good.
Neuroimaging predictors of iTBS response to treatment - Well-being (WEMWBS) | 6 week
  For secondary analyses, improvement in symptoms will be defined as the percentage of change of symptoms at week 6 in comparison with pre-treatment symptoms severity. Response to treatment will be defined as a 50% reduction in pre-treatment symptoms severity. The Short Warwick Edinburgh Mental Well-Being Scale (SWEMWBS) will be used to assess general overview of mental well-being. It's a self-rated; 7 questions; rated over the past 2 weeks. Scored: 1 (none of the time) to 5 (all of the time).

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tremblay, PhD, Principal Investigator — The Royal Ottawa Mental Health Centre
Locations (1):
- The Royal Ottawa Mental Health Centre, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All Individual Participant Data collected from this study (IPD) will be de-identified for all parties who have permission to access it. This de-identified data may be shared with other researchers at the Royal's Institute of Mental Health Research. De-identified may be shared with the public only upon request. Please note that all data that has the potential of revealing participants' identity will NOT be used to shared.
Time Frame: De-identified data may become available (upon request) when the study is completed and published (anticipated time frame: the year of 2024)
Access Criteria: De-identified data will be accessible only through the permission of the lead research scientist. All requests must be made and accepted by her.